CLINICAL TRIAL: NCT02255552
Title: An Open-Label, Multi-Center, Study With a Concurrent Untreated Control Arm to Evaluate the Efficacy and Safety of Eteplirsen in Duchenne Muscular Dystrophy
Brief Title: Study of Eteplirsen in DMD Patients
Acronym: PROMOVI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4658-301
Record Dates: First submitted 2014-09-25; First posted 2014-10-02 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-12

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: DMD, Duchenne, Eteplirsen, dystrophy, dystrophin, exon 51
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — eteplirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treated Group (Experimental): Approximately 80 patients with genotypically confirmed Duchenne muscular dystrophy (DMD) with genetic deletions amenable to treatment by exon 51 skipping will receive 30 mg/kg of eteplirsen weekly for 96 weeks, followed by a safety extension (not to exceed 48 weeks).
  Interventions: Drug: eteplirsen
- Untreated Group (No Intervention): Approximately 30 DMD patients not amenable to exon 51 skipping will not receive eteplirsen.

INTERVENTIONS:
Drug: eteplirsen — Eteplirsen 30 mg/kg will be administered as an IV infusion once a week for 96 weeks, followed by a safety extension (not to exceed 48 weeks).
  Other Names: AVI-4658; EXONDYS 51®
  Arms: Treated Group

SUMMARY:
The main objective of this study is to provide evidence of efficacy of eteplirsen (AVI-4658) in Duchenne muscular dystrophy (DMD) patients that are amenable to skipping exon 51. Additional objectives include evaluation of safety, biomarkers and the long-term effects of eteplirsen up to 96 weeks, followed by a safety extension (not to exceed 48 weeks).

DETAILED DESCRIPTION:
This is an open-label, multi-center study to evaluate the efficacy and safety of eteplirsen in patients with genotypically confirmed Duchenne muscular dystrophy (DMD) with genetic deletions amenable to exon 51 skipping (treated group), with a concurrent control arm of DMD patients not amenable to exon 51 skipping (untreated group). Following primary efficacy endpoints, dosing will continue to week 144 to evaluate the long term effects of eteplirsen.

Patients in the treated group will receive once weekly intravenous (IV) infusions of 30 mg/kg Eteplirsen for 96 weeks, followed by a safety extension (not to exceed 48 weeks). Patients in the untreated group will not receive treatment.

Clinical efficacy will be assessed at regularly scheduled study visits, including functional tests such as the six minute walk test. Patients in the treated group will undergo a muscle biopsy at Baseline and a second muscle biopsy over the course of the study. Patients in the untreated group will not undergo muscle biopsy.

Safety, including adverse event monitoring and routine laboratory assessments, will be continuously monitored for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Male 7-16 years old
* Diagnosed with DMD, genotypically confirmed
* Stable dose of corticosteroids for at least 24 weeks
* Have intact right and left alternative upper muscle groups
* Mean 6MWT greater than 300m (primary analysis on 300 to 450 meters)
* Stable pulmonary and cardiac function: predicted FVC equal to or greater than 50% and LVEF of greater than 50%

Exclusion Criteria:

* Previous treatment with drisapersen or any other RNA antisense agent or any gene therapy within the last 6 months
* Participation in any other DMD interventional clinical study within 12 weeks
* Major surgery within 3 months
* Presence of other clinically significant illness
* Major change in the physical therapy regime within 3 months

Other inclusion/exclusion criteria apply.

Ages: 7 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (37):
- United States (37):
  - Neuromuscular Research Center, Phoenix, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - Rady Children's Hospital, U.C. San Diego, San Diego, California
  - Stanford University School of Medicine/Medical Center, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Health System, Washington D.C., District of Columbia
  - The University of Florida, Powell Gene Therapy Center, Gainesville, Florida
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Rare Disease Research Center, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - University of Rochester Clinical Research Center, Rochester, New York
  - Levine Childrens Hospital, Carolinas Medical Center, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center (CCHMC), Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Shriners Hospital for Children, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brogna C, Coratti G, Pane M, Ricotti V, Messina S, D'Amico A, Bruno C, Vita G, Berardinelli A, Mazzone E, Magri F, Ricci F, Mongini T, Battini R, Bello L, Pegoraro E, Baranello G, Previtali SC, Politano L, Comi GP, Sansone VA, Donati A, Bertini E, Muntoni F, Goemans N, Mercuri E; on behalf on the International DMD group. Long-term natural history data in Duchenne muscular dystrophy ambulant patients with mutations amenable to skip exons 44, 45, 51 and 53. PLoS One. 2019 Jun 25;14(6):e0218683. doi: 10.1371/journal.pone.0218683. eCollection 2019. PMID 31237898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 40 sites in the United States.
Pre-assignment Details: A total of 109 participants were enrolled in the study. Only 79 participants were treated and the remaining participants were not applicable for treatment as those participants assessed under "Untreated" arm.
Groups:
- Eteplirsen 30 mg/kg: Participants with genotypically confirmed Duchenne muscular dystrophy (DMD) with genetic deletions amenable to treatment by exon 51 skipping received Eteplirsen as an Intravenous (IV) infusion, at a dose of 30 milligram per kilogram (mg/kg) once weekly for 96 weeks.
- Untreated Control Group (Non-exon 51 Amenable Participants): DMD participants with mutations amenable to skipping of any exon(s) except exon 51 did not receive any treatment, but completed study assessments up to 96 weeks.
Period: Overall Study
Arm/Group | Eteplirsen 30 mg/kg | Untreated Control Group (Non-exon 51 Amenable Participants)
Started | 79 | 30
Completed | 78 | 15
Not Completed | 1 | 15
Not completed — Participants enrolled into another study | 0 | 11
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Population: Consisted of all participants who received at least 1 dose of eteplirsen in the eteplirsen-treated group or had at least 1 post-baseline safety assessment in the untreated group.Comparisons between the eteplirsen-treated and the untreated group were not to be performed due to the small number of subjects and differences in the population groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eteplirsen 30 mg/kg | Untreated Control Group (Non-exon 51 Amenable Participants) | Total
Number analyzed (Participants) | 79 | 30 | 109
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.1 (2.04) | 8.8 (1.76) | 9.0 (1.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 79 | 30 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 71 | 24 | 95
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 2 | 0 | 2
  White | 67 | 26 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 79 | 30 | 109

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 6 Minute Walk Test (6MWT) Distance at Week 96
Description: 6MWT was performed by standardized procedures for all participants. Participants were asked to walk a set course of 25 meters for 6 minutes (timed), and the distance walked (in meters) was recorded. Change from baseline in 6MWT distance at Week 96 was reported.
Time Frame: Baseline, Week 96
Population: Primary efficacy set: all participants in the efficacy set (all participants in eteplirsen-treated and untreated control groups who had at least 1 post-baseline functional assessment) who had a Baseline 6MWT distance of 300 to 450 meters, inclusive. Here, "Overall Number of Participants Analyzed"=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Eteplirsen 30 mg/kg | Untreated Control Group (Non-exon 51 Amenable Participants)
Number analyzed (Participants) | 65 | 9
meters | -117.91 (128.488) | -133.56 (129.333)

2. Secondary Outcome: Change From Baseline in Dystrophin Protein Levels Determined by Western Blot at Week 96
Description: Change from baseline in dystrophin protein levels (in muscle biopsy samples) were determined by Western blot. For each time point, 2 blocks of tissues were analyzed by Western blot, each with 2 replicates of gels to determine the dystrophin level as compared to a healthy individual (Percent Normal). The block average value from 2 replicate gels was computed. The overall average was calculated as the mean of the block average values. The overall average values were used for all analyses. In case only 1 gel was available for a block, then that value was used as the block average value.
Time Frame: Baseline, Week 96
Population: Analysis Set consisted of a subset of participants who received at least 1 dose of eteplirsen and had both baseline and 1 post-dose muscle biopsy samples evaluable for dystrophin expression at Week 96. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for the Untreated Control group.
Measure: Mean (Standard Deviation); unit: Percent Normal Dystrophin Protein Level
Arm/Group | Eteplirsen 30 mg/kg
Number analyzed (Participants) | 16
Percent Normal Dystrophin Protein Level | 0.516 (0.7236)

3. Secondary Outcome: Number of Participants Having Ability to Rise Independently From the Floor Determined Based on North Star Ambulatory Assessment (NSAA) at Week 96
Description: NSAA is a clinician-administered scale that rates participant performance on 17-items and included assessments of abilities such as 10-meter walk/run, rising from a sit to stand, standing on 1 leg, climbing a box step, descending a box step, rising from lying to sitting, rising from the floor, lifting the head, standing on heels, and jumping. For all activities, participants were graded as follows: 0 = unable to achieve goal independently; 1 = modified method but achieves goal independent of physical assistance from another and 2 = normal, no obvious modification of activity. Number of participants having ability to rise independently from the floor indicated by a NSAA Rise from floor sub score greater than 0 (unable to achieve goal independently) was reported.
Time Frame: Week 96
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg | Untreated Control Group (Non-exon 51 Amenable Participants)
Number analyzed (Participants) | 61 | 9
Participants | 33 | 3

4. Secondary Outcome: Number of Participants Who Lost Ambulation (LOA) by Week 96
Description: Number of participants who lost ambulation (LOA) by Week 96 was reported. Participant were considered non-ambulatory if each of the 3 conditions below were met: NSAA walk subscore was "0" (unable to achieve goal independently) on 2 consecutive days within a visit or NSAA was not done due to reason related to non-ambulation; 6MWT was not done with any reason related to permanent non-ambulation; and no later data showing this participant was still ambulatory. This was not required if non ambulatory status occurred at the time of early withdrawal or at the end of Week 96 assessment. NSAA is a 17-item scale to assess the participant's abilities; total score range from 0 (if all the activities are failed) to 34 (if all the activities are achieved) with higher scores indicating better performance on the assessment/ fully-independent function.
Time Frame: Up to Week 96
Population: Primary efficacy set consisted of all participants in the efficacy set (all participants in eteplirsen-treated and untreated control groups who had at least 1 post-baseline functional assessment) who had a Baseline 6MWT distance of 300 to 450 meters, inclusive.
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg | Untreated Control Group (Non-exon 51 Amenable Participants)
Number analyzed (Participants) | 67 | 20
Participants | 12 | 1

5. Secondary Outcome: Change From Baseline in Forced Vital Capacity Percent (FVC%) Predicted at Weeks 96
Description: FVC is the total amount of air exhaled during the forced expiratory volume test that is measured during spirometry; and is the most important measurement of lung function. This test requires participant to breath into a tube connected to a machine that measures the amount of air that can be moved in and out of the lungs after taking an inhaled bronchodilator medicine which is used to dilate participant's bronchial (breathing) tubes. Percent of predicted FVC = (observed value) / (predicted value) * 100%.
Time Frame: Baseline, Week 96
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of predicted FVC
Arm/Group | Eteplirsen 30 mg/kg | Untreated Control Group (Non-exon 51 Amenable Participants)
Number analyzed (Participants) | 66 | 9
Percentage of predicted FVC | -3.413 (12.4011) | -2.461 (9.6000)

6. Secondary Outcome: Change From Baseline in North Star Ambulatory Assessment (NSAA) Total Scores at Week 96
Description: NSAA is a clinician-administered scale that rates participant performance on 17-items and included assessments of abilities such as 10-meter walk/run, rising from a sit to stand, standing on 1 leg, climbing a box step, descending a box step, rising from lying to sitting, rising from the floor, lifting the head, standing on heels, and jumping. Participant were graded as follows: 0 = unable to achieve goal independently; 1 = modified method but achieves goal independent of physical assistance from another and 2 = normal, no obvious modification of activity. NSAA total score was derived by summing the scores for all the individual items and range from 0 (if all the activities are failed) to 34 (if all the activities are achieved) with higher scores indicating better performance on the assessment/ fully-independent function.
Time Frame: Baseline, Week 96
Population: Primary efficacy: all participants in the efficacy set (all participants in eteplirsen-treated and untreated control groups who had at least 1 post-baseline functional assessment) who had a Baseline 6MWT distance of 300 to 450 meters, inclusive. Here, "Overall Number of Participants Analyzed"=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Eteplirsen 30 mg/kg | Untreated Control Group (Non-exon 51 Amenable Participants)
Number analyzed (Participants) | 61 | 9
Unit on scale | -7.23 (5.173) | -8.44 (9.812)

7. Secondary Outcome: Change From Baseline in Dystrophin Intensity Levels Determined by Immunohistochemistry (IHC) at Week 96
Description: Change from baseline in dystrophin intensity levels (in muscle biopsy samples) was determined by Immunohistochemistry.
Time Frame: Baseline, Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent dystrophin positive fibers
Arm/Group | Eteplirsen 30 mg/kg
Number analyzed (Participants) | 16
Percent dystrophin positive fibers | 0.030 (0.0360)

ADVERSE EVENTS:
Time Frame: From start of study drug administration to Week 144
Arm/Group | Eteplirsen 30 mg/kg | Untreated Control Group (Non-exon 51 Amenable Participants)
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/30
Serious Adverse Events (participants affected / at risk) | 11/79 | 2/30
Other Adverse Events (participants affected / at risk) | 78/79 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eteplirsen 30 mg/kg (N=79) | Untreated Control Group (Non-exon 51 Amenable Participants) (N=30)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Abasia (General disorders) | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Lymphadenitis viral (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eteplirsen 30 mg/kg (N=79) | Untreated Control Group (Non-exon 51 Amenable Participants) (N=30)
Flushing (Vascular disorders) | 4 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Seasonal allergy (Immune system disorders) | 14 | 0
Pyrexia (General disorders) | 20 | 1
Non-cardiac chest pain (General disorders) | 9 | 0
Fatigue (General disorders) | 8 | 0
Catheter site pain (General disorders) | 7 | 0
Peripheral swelling (General disorders) | 5 | 0
Infusion site bruising (General disorders) | 4 | 0
Infusion site pain (General disorders) | 4 | 0
Anxiety (Psychiatric disorders) | 6 | 1
Insomnia (Psychiatric disorders) | 4 | 0
Procedural pain (Injury, poisoning and procedural complications) | 25 | 0
Contusion (Injury, poisoning and procedural complications) | 24 | 1
Fall (Injury, poisoning and procedural complications) | 22 | 6
Skin abrasion (Injury, poisoning and procedural complications) | 21 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 12 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 10 | 1
Muscle strain (Injury, poisoning and procedural complications) | 7 | 0
Laceration (Injury, poisoning and procedural complications) | 4 | 1
Limb injury (Injury, poisoning and procedural complications) | 4 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 | 0
Torus fracture (Injury, poisoning and procedural complications) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 25 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 22 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Headache (Nervous system disorders) | 40 | 1
Dizziness (Nervous system disorders) | 9 | 0
Migraine (Nervous system disorders) | 4 | 0
Ear pain (Ear and labyrinth disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 39 | 0
Diarrhoea (Gastrointestinal disorders) | 20 | 1
Nausea (Gastrointestinal disorders) | 17 | 0
Abdominal pain upper (Gastrointestinal disorders) | 14 | 3
Abdominal pain (Gastrointestinal disorders) | 8 | 0
Constipation (Gastrointestinal disorders) | 8 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 1
Abdominal discomfort (Gastrointestinal disorders) | 4 | 1
Proteinuria (Renal and urinary disorders) | 8 | 0
Rash (Skin and subcutaneous tissue disorders) | 17 | 2
Erythema (Skin and subcutaneous tissue disorders) | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 2
Nasopharyngitis (Infections and infestations) | 29 | 3
Upper respiratory tract infection (Infections and infestations) | 25 | 1
Ear infection (Infections and infestations) | 11 | 0
Influenza (Infections and infestations) | 8 | 1
Gastroenteritis (Infections and infestations) | 7 | 1
Gastroenteritis viral (Infections and infestations) | 7 | 0
Pharyngitis streptococcal (Infections and infestations) | 6 | 1
Sinusitis (Infections and infestations) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT02255552/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT02255552/SAP_001.pdf